CLINICAL TRIAL: NCT02130375
Title: Clinical and Urodynamic Effects of Minimally Laser (IncontiLaseTM) Procedure for Female Stress Urinary Incontinence
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201402021RINB
Record Dates: First submitted 2014-04-28; First posted 2014-05-05 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2016-01

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- stress urinary incontinence (Experimental): Women with stress urinary incontinence
  Interventions: Procedure: the IncontiLaseTM procedure

INTERVENTIONS:
Procedure: the IncontiLaseTM procedure — Utilizing laser (IncontiLaseTM) to treat the anterior vaginal wall area to intensify periurethral tissue and achieve urinary continence

SUMMARY:
The purpose of this study is to get the effect of IncontiLaseTM procedure; and its impact on urinary symptoms and female sexual function.

DETAILED DESCRIPTION:
To get the objective urodynamic and sonographic effects of IncontiLaseTM procedure on women with stress urinary incontinence; and its impact on urinary symptoms and female sexual function.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive sexually active and parous adult women with the complaint of stress urinary incontinence

Exclusion Criteria:

* < 20 years old female

Ages: 20 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2014-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
The change of pad weight from baseline | 3 months
  The change of pad weight from baseline after IncontiLaseTM procedure

SECONDARY OUTCOMES:
The change of maximum urethral closure procedure from baseline | 3 months
  The change of maximum urethral closure procedure from baseline after the IncontiLaseTM procedure by urodynamic studies

OTHER OUTCOMES:
The change of female sexual functional score from baseline after treatment | 3 months
  The change of female sexual functional score from baseline after treatment
The change of periurethral blood flow from baseline | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Ho-Hsiung Lin, MD, PhD, Principal Investigator — Department of Obstetrics & Gynecology, National Taiwan University Hospital
Locations (1):
- Department of Obstetrics & Gynecology, National Taiwan University Hospital, Taipei, Taiwan